CLINICAL TRIAL: NCT00526253
Title: A Multicenter Study to Assess the Safety and Cardiovascular Effects of Myocell™ Implantation by a Catheter Delivery System in Congestive Heart Failure Patients Post Myocardial Infarction(s)
Brief Title: To Assess Safety and Efficacy of Myoblast Implantation Into Myocardium Post Myocardial Infarction
Acronym: MARVEL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioheart, Inc. (Industry)
Responsible Party: Warren Sherman, MN, Center for Interventional Vascular Therapy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMI-WW-02-003
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; CHF; Heart Disease; Heart Attack; Stem Cell; Myoblast; Bioheart
MeSH Terms: conditions — Heart Failure; Heart Diseases; Myocardial Infarction | interventions — hypothermosol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Active Comparator): Patient will undergo biopsy. Skeletal myoblasts will be cultured in growth media.
  Interventions: Biological: MyoCell
- High Dose (Active Comparator): Patient will undergo biopsy. Skeletal myoblasts will be cultured in growth media.
  Interventions: Biological: MyoCell
- Control (Placebo Comparator): Patient will undergo biopsy of muscle tissue and biopsy tissue will be sent to lab.
  Interventions: Procedure: Hypothermosol

INTERVENTIONS:
Biological: MyoCell — Patient will receive injections of cultured, expanded skeletal myoblasts into the myocardium at a dose of 400 million cells.
  Arms: Low Dose
Biological: MyoCell — Patient will receive injections of cultured, expanded skeletal myoblasts into the myocardium at a dose of 800 million cells.
  Arms: High Dose
Procedure: Hypothermosol — After the cell culture period of time has passed, patient's myocardium will be injected with the transport media alone. Patient will not receive any cultured myoblasts during these injections.
  Arms: Control

SUMMARY:
This study injects a person's own stem cells into heart muscle tissue after a person has one or more heart attacks. The purpose of the study is whether the stem cells will improve a patient's heart performance.

DETAILED DESCRIPTION:
Autologous myoblasts are harvested from a patient's skeletal muscle tissue. The myoblasts are isolated and expanded in culture in a closed system. When a sufficient number of cells are estimated they are taken from culture, packaged in a suspension and sent to the patient's interventionalist. The interventionalist uses an injection catheter via femoral artery to inject the myoblasts directly into the myocardium.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet ALL of the following inclusion criteria during the screening/enrollment visit #1 and prior to being randomized into the study. Screening/enrollment visit #1 is defined to start the date the ICF is signed by the patient:

1. Chronic CHF, New York Heart Association (NYHA) Class II-IV;
2. Stable and on optimal medical management for greater or equal to 60 days as follows:

   1. systolic and diastolic hypertension controlled in accordance with contemporary guidelines;
   2. patient stabilized on maximum tolerated dose of beta blockers;
   3. patient stabilized on maximum tolerated dose of angiotensin concerting enzyme (ACE) inhibitors;
   4. patients intolerant of ACE inhibitors should be stabilized on angiotensin receptor blockers (ARB);
   5. fluid control with diuretics and a salt restricted diet;
   6. patients with sever symptoms of heart failure (Class III-IV) lacking contraindications to aldosterone antagonism and not on both ACE inhibitors and ARBs have been considered for such therapy.
3. Age 18-80;
4. Left ventricular ejection fraction (LVEF) at screening of less than or equal to 35 percent by multiple gaited acquisition scan (MUGA);
5. Need or feasibility for revascularization has been ruled out by previous coronary angiogram or ruled out to the satisfaction of the investigator via previous conventional stress study completed within 1 year of screening. The need or feasibility for revascularization will be reassessed at screening using dobutamine stress echocardiography (DSE);
6. Defined region of mycardial dysfunction related to previous MI involving the anterior, later, posterior or inferior walls including the apical septum (excluding the basal septum) assessed by a large area of akinesia in the left ventricle (using DSE at screening);
7. B-type natriuretic peptide (BNP) or NT pro-BNP is above the upper limit of normal.

Exclusion Criteria:

1. Non-pregnant women who are not postmenopausal, surgically sterile or not practicing an acceptable method of contraception. A female patient of child bearing potential, with a positive serum or urine pregnancy test at screening visit #1. Females refusing to exercise a reliable form of contraception;
2. Myocardial wall thickness of <6 mm (millimeters) in the akinetic myocardial region to be injected (using DSE at screening)
3. Inability to undergo a surgical biopsy of the skeletal muscle for culture of myoblasts, including any significant myopathy;
4. Patient will require revascularization within six months;
5. Patients on continuous or intermittent intravenous drug therapy;
6. Not fitted, or fitted within less than 90 days prior to screening visit #1, with an implantable cardioverter defibrillator (ICD);
7. Sustained ventricular tachycardia (VT), automatic implantable cardiodefibrillator (AICD) firing, or ventricular fibrillation (VF) within 90 days prior to screening visit #1;
8. Inability to perform a 6 minute walk test due to physical limitations other than HF including:

   1. Severe peripheral vascular disease, including aortic aneurysms, leading to limited claudication;
   2. Severe pulmonary disease or chronic obstructive pulmonary disease (COPD) limiting exercise, dependence on chronic oral steroid therapy or previously requiring mechanical ventilation;
   3. Stroke or transient ischemic attack leading to limitations in lower extremities or occurring within 180 days prior to screening visit #1;
9. MI, unstable angina or percutaneous coronary intervention (PCI) within 90 days prior to screening;
10. having undergone CABG surgery within 150 days prior to screening visit #1;
11. Active myocarditis, constrictive pericarditis, restrictive, hypertrophic or congenital cardiomyopathy;
12. Hemodynamically significant severe primary valvular heart disease, unless corrected by a properly functional prosthetic valve;
13. Prior aortic valve replacement;
14. Systolic blood pressure (supine) ≤90 mmHg;
15. Resting heart rate >100 bpm;
16. Severe uncontrolled HF including any evidence of severe fluid overload such as peripheral edema >+2 or rales ≥1/3 the lungs' height, need for intravenous therapy for HF within 60 days of screening visit #1 or hospitalization for HF within 90 days of screening visit #1;
17. Patient scheduled to receive cardiac resynchronization therapy (CRT) during the study;
18. Expected to receive or received a cardiac transplant, surgical remodeling procedure, left ventricular assist device or cardiomyoplasty;
19. Six-minute walk test (6MWT) of >400 meters or Minnesota Living With Heart Failure (MLWHF) score of <20;
20. Hematocrit (HCT) concentration below 30% (males) or below 27% (females);
21. Serum creatinine greater than 2.5 mg/dL (milligrams per deciliter) or end stage renal disease;
22. Left ventricular mural thrombus;
23. Known sensitivity to gentamicin sulfate; or severe adverse reaction to nonionic radiocontrast agents;
24. Active infectious disease and/or known to have tested positive for human immunodeficiency virus (HIV), human t lymphotrophic virus (HTLV), hepatitis B virus (HBV), hepatitis C virus (HCV), cytomegalovirus (CMV); immunoglobulin M [IgM], and/or syphilis. If the panel includes antibodies to the HBV core antigen (HBV-cAg) and hepatitis B surface antigen (HBV-sAg), then an expert will be consulted as to patient's eligibility based on the patient's infectious status;
25. Patients have undergone enhanced external pulsation (EECP) tratment within the last 6 months;
26. Exposure to any previous experimental angiogenic therapy and/or myocardial laser therapy, or therapy with another investigational drug within 60 days of screening visit #1 or enrollment in any concurrent study that may confound the results of this study;
27. Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
28. Any illness other than CHF which might reduce life expectancy to less than 1 year from screening visit #1;
29. Recent initiation of cardiac resynchronization therapy via placement of a bi-ventricular pacemaker or bi-ventricular AICD within 180 days of study enrollment; and

30 Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2007-09; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | 6 months
Quality of Life Questionnaire | 6 months

SECONDARY OUTCOMES:
Hospitalization occurrences | 12 months

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Cardiology, P.C., Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Arizona Heart Institute, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scripps Green Hospital, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Jim Moran Heart and Vascular Research Institute, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida Shands, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Florida Hospital Center Cardiovascular Center, Orlando, Florida
  - Emory/Crawford Long, Atlanta, Georgia
  - St. Joseph's Research Institute/ACRI, Atlanta, Georgia
  - RUSH University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Gagnon Heart Hospital, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Center, Cincinnati, Ohio
  - University Hospital, Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Stern Cardiology, Germantown, Tennessee
  - Texas Heart Institute, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- See also: Bioheart Inc. website — http://www.bioheartinc.com